CLINICAL TRIAL: NCT07125456
Title: The Effect of Simulation-Based Learning Experiences on Nursing Students' Knowledge, Skills and Self-Efficacy Levels in Teaching Postmortem Care
Brief Title: The Effect of Simulation-Based Postmortem Care on Nursing Students' Knowledge, Skills, and Self-Efficacy Levels
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Ozan Acar, Principal Investigator, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2025-12/453
Record Dates: First submitted 2025-08-05; First posted 2025-08-15 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Postmortem Care
Keywords: Postmortem Changes; High Fidelity Simulation Nursing; Nursing Students; Knowledge; Nursing Care; Self-Efficacy; Education, Nursing
MeSH Terms: conditions — Postmortem Changes

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Postmortem Care Simulation (Experimental): Postmortem Care Teaching Simulation
  Interventions: Other: Postmortem Care Teaching Simulation
- Traditional Education Arm (No Intervention): Theoretical Postmortem Care Education and Postmortem Care Skills Video

INTERVENTIONS:
Other: Postmortem Care Teaching Simulation — The participants in the experimental group will be administered the "Informed Consent Form," "Demographic Characteristics Form," "Postmortem Care Knowledge Test for Nursing Students (PCKTNS)," and "End-of-Life and Postmortem Care Self-Efficacy Scale for Nursing Students (ELPMCSESN)" prior to the theoretical education. Following the pre-tests, it is planned to provide theoretical education for approximately 4 class hours (with each class hour lasting 45 minutes). The first 2 hours of the theoretical education will cover topics related to Death and General Aspects of Death, while the remaining 2 class hours will be delivered as a PowerPoint presentation focusing on postmortem care application content.
  Following the theoretical education, the experimental and control groups will be shown the "Postmortem Care Skills Video." Additionally, prior to the teaching simulation for postmortem care, the experimental group will be shown the "Scenario Case Video," after which the scenario prepared fo
  Arms: Postmortem Care Simulation

SUMMARY:
PURPOSE AND TYPE OF THE RESEARCH This study is designed as a randomized controlled experimental study to investigate the impact of simulation-based learning experiences in the teaching of postmortem care on the knowledge, skills, and self-efficacy levels of nursing students.

RESEARCH HYPOTHESES

Hypothesis 1 (H1): The postmortem care knowledge levels of students who experience simulation-based learning are higher compared to those taught through traditional methods.

Hypothesis 2 (H2): The postmortem care skill levels of students who experience simulation-based learning are higher compared to those taught through traditional methods.

Hypothesis 3 (H3): The self-efficacy levels of students who experience simulation-based learning in end-of-life and postmortem care are higher compared to those taught through traditional methods.

Additionally, it is anticipated that students who undergo simulation-based learning experiences will exhibit higher levels of student satisfaction and confidence in their learning process within this study.

DETAILED DESCRIPTION:
The purpose of nursing is to provide individualized care to meet the needs of an individual throughout their lifespan, which begins with fertilization and ends with death. In alignment with this fundamental objective, nurses facilitate the preservation, maintenance, and enhancement of an individual's health, the restoration of function or recovery in cases of illness, and the provision of a peaceful, dignified, and good death during the final stages of life. The end-of-life period is defined as the individual's last months and days. End-of-life care encompasses a comprehensive approach that includes appropriate nursing interventions addressing the bio-physiological, psychological, social, cultural, and environmental dimensions of an individual before, during, and after death (postmortem). This form of care serves as an indicator of the quality of patient care and assists family members in accepting the reality of death through family-centered approaches. The final phase of end-of-life care, postmortem care, holds significant importance as it involves the nurse's awareness of their own emotions, the preservation of the deceased individual's dignity until the very end, the provision of opportunities for family members or loved ones to initiate a positive grieving process through farewell and religious/cultural rituals, and the fulfillment of legal and procedural requirements. Postmortem care entails the physical care of the deceased individual, delivered in a manner respectful of the values and preferences of both the deceased and their family members, while adhering to infection control measures, ethical standards, and legal protocols. Additionally, it includes the provision of psychosocial support to grieving family members during the mourning process. Despite its critical role within palliative care in nursing, there is a notable scarcity of research focused on postmortem care. Death represents the final stage of life, a universal experience for all living organisms, marking the irreversible cessation of vital functions. According to the World Health Organization (WHO) 2024 statistics, approximately 60 million individuals die globally each year, equating to an average of 164,000 deaths per day. Historically, death frequently occurred in home settings; however, the increasing and aging population, the rise in chronic diseases, and advancements in medical diagnostics, care, and treatment interventions that extend life have led to the hospitalization of terminally ill individuals for ongoing care and treatment. These factors have resulted in the majority of deaths occurring in healthcare settings, such as hospitals, thereby increasing the likelihood of nurses and nursing students encountering death. Studies involving nursing students have highlighted that providing care to individuals in the dying process, those nearing death, or the deceased presents multifaceted challenges and is considered a significant issue. Previous research has indicated that nursing students' initial experiences with patient death are often accompanied by negative emotions such as fear, sadness, disappointment, anxiety, helplessness, inadequacy, and guilt. Furthermore, these emotions may lead nursing students to adopt maladaptive coping mechanisms, including suppression, avoidance, and detachment. Limited studies related to this topic have revealed that nursing students feel inadequately prepared and struggle to cope with death and postmortem care, reporting a lack of readiness to care for the deceased and their families. In Turkey, limited descriptive and qualitative studies with nursing students have identified deficiencies in knowledge regarding end-of-life care, as well as difficulties in managing and delivering such care. However, it is imperative that nursing students possess adequate knowledge and skills to address challenging situations, such as postmortem care. Moreover, their self-efficacy levels are critical in effectively applying these knowledge and skills. The concept of self-efficacy reflects the distinction between possessing knowledge and skills and utilizing these abilities in challenging contexts. Consequently, education and training play a pivotal role in fostering knowledge, skills, and self-efficacy in end-of-life and postmortem care. Nevertheless, global undergraduate nursing curricula are noted for their deficiencies in addressing end-of-life and postmortem care education and a strong emphasis is placed on the need for enhanced training at the undergraduate level. Studies further indicate that postmortem care education is inadequately addressed, with students feeling unprepared and exhibiting low self-efficacy in providing postmortem care. Such education is often limited to theoretical discussions within the broader context of end-of-life or palliative care. A review of international literature reveals only one non-randomized pre-test/post-test study implementing an augmented reality-based mentorship program for newly graduated nurses in postmortem care. Similarly, a national literature review identified a single study by Uzun and Cerit (2024) that utilized creative drama to deliver postmortem care education to nursing students. These studies suggest that augmented reality and creative drama methods effectively enhance postmortem knowledge and skills; however, they underscore the need for further research, particularly randomized controlled trials. Additionally, while self-efficacy-a factor potentially influencing students' readiness for end-of-life care-has been explored in non-experimental studies, no studies have specifically addressed it in the context of postmortem care. A comprehensive review, however, suggests that simulation-based learning methods in nursing education could address the educational needs in end-of-life and postmortem care. The literature further recommends that simulation methods be employed, as they are considered an effective means of developing skills expected of all nurses in end-of-life care. Simulation-based learning is defined as a learning process that replicates situations or events as closely as possible to those encountered in clinical practice. Increasingly utilized in nursing education over the years, this method provides nursing students with safe environments to practice and enhance their skills. Simulation-based learning offers a secure setting, particularly in hospitals and other care delivery environments, to address complex challenges such as sudden changes in a patient's condition or the care of multiple patients. It enables healthcare professionals to minimize the risk of patient harm while ensuring the provision of adequate and high-quality care. Studies suggest that simulations related to end-of-life care can positively influence nursing students' knowledge, confidence, and communication skills, although the number of such simulation studies remains limited, indicating a need for further research. However, no studies have been identified that utilize high-fidelity simulation as a method to acquire competencies (knowledge, skills, and self-efficacy) in end-of-life and postmortem care. This research aims to determine the impact of simulation-based learning experiences on the knowledge, skills, and self-efficacy levels of nursing students in the teaching of postmortem care.

ELIGIBILITY:
Inclusion Criteria:

* Be literate in Turkish
* Be 18 years of age or older
* Have no history of or current psychiatric disorders/illnesses, not be undergoing any psychiatric treatment, and not be taking any psychiatric medication
* Not have previously taken any training or courses in postmortem care
* Not have previously provided postmortem care.

Exclusion Criteria:

* Losing a loved one within the last year

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2025-11-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Postmortem Care Skills | Average postmortem care skill level in 1 month
  Following the theoretical education, both the experimental and control groups will be shown the "Postmortem Care Skills Video." Additionally, prior to the teaching simulation for postmortem care, the experimental group will be shown the "Scenario Case Video," after which the scenario prepared for the teaching simulation will be implemented. At this stage, no intervention will be applied to the control group. Four weeks after the learning simulation administered to the experimental group, participants from both the experimental and control groups will be taken to the evaluation simulation in pairs. Prior to the postmortem care evaluation simulation, students from both the experimental and control groups will be shown the "Scenario Case Video," followed by the application of the scenario prepared for the evaluation simulation. At this stage, participants will be evaluated according to the "Postmortem Care Simulation Checklist." Following the evaluation simulation, the students will be a
Postmortem Care Simulation - Assessment Simulation | Changes in postmortem care skills one month after postmortem care simulation
  Following the theoretical education, both the experimental and control groups will be shown the "Postmortem Care Skills Video." Additionally, prior to the teaching simulation for postmortem care, the experimental group will be shown the "Scenario Case Video," after which the scenario prepared for the teaching simulation will be implemented. At this stage, no intervention will be applied to the control group. Four weeks after the learning simulation administered to the experimental group, participants from both the experimental and control groups will be taken to the evaluation simulation in pairs. Prior to the postmortem care evaluation simulation, students from both the experimental and control groups will be shown the "Scenario Case Video," followed by the application of the scenario prepared for the evaluation simulation. At this stage, participants will be evaluated according to the "Postmortem Care Simulation Checklist." Following the evaluation simulation, the students will be a

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared, as informed consent for data sharing has not yet been obtained from participants. This decision aligns with current ethical guidelines and is subject to future approval by the ethics committee.

REFERENCES:
- [Result] Uzun, L. N. (2023). The effect of the creative drama method on the knowledge, skills, and satisfaction of nursing students regarding postmortem care (Doctoral dissertation, Bolu Abant İzzet Baysal University, Graduate School of Education, Department of Nursing).
- [Result] Unver V, Basak T, Watts P, Gaioso V, Moss J, Tastan S, Iyigun E, Tosun N. The reliability and validity of three questionnaires: The Student Satisfaction and Self-Confidence in Learning Scale, Simulation Design Scale, and Educational Practices Questionnaire. Contemp Nurse. 2017 Feb;53(1):60-74. doi: 10.1080/10376178.2017.1282319. Epub 2017 Feb 10. PMID 28084900
- [Result] Tamaki T, Inumaru A, Yokoi Y, Fujii M, Tomita M, Inoue Y, Kido M, Ohno Y, Tsujikawa M. The effectiveness of end-of-life care simulation in undergraduate nursing education: A randomized controlled trial. Nurse Educ Today. 2019 May;76:1-7. doi: 10.1016/j.nedt.2019.01.005. Epub 2019 Jan 27. PMID 30738199
- [Result] Roberts, D. (2019). Dying. In K. Holland & J. Jenkins (Eds.), Applying the Roper-Logan-Tierney model in practice (3rd ed., pp. 453-472). Elsevier. https://doi.org/10.1016/B978-0-7020-4658-2.00014-4
- [Result] Rattani SA, Kurji Z, Khowaja AA, Dias JM, AliSher AN. Effectiveness of High-Fidelity Simulation in Nursing Education for End-of-Life Care: A Quasi-experimental Design. Indian J Palliat Care. 2020 Jul-Sep;26(3):312-318. doi: 10.4103/IJPC.IJPC_157_19. Epub 2020 Aug 29. PMID 33311872
- [Result] Perry, A. G., Potter, P. A., Ostendorf, W. R., & Laplante, N. (2025). End-of-life care. In A. G. Perry, P. A. Potter, W. R. Ostendorf, & N. Laplante (Eds.), Clinical nursing skills and techniques (11th ed., pp. 498-518). Elsevier. https://doi.org/10.1016/B978-0-443-10718-4.00026-0
- [Result] Karakurt, P. (2024). Loss and the death process. In T. Atabek Aştı & A. Karadağ (Eds.), Fundamentals of nursing: From knowledge to practice: Concepts - principles - skills (Updated and expanded 3rd ed., Vol. 2, pp. 983-998). İstanbul: Akademi Basın ve Yayıncılık.
- [Result] Jeffries PR. A framework for designing, implementing, and evaluating simulations used as teaching strategies in nursing. Nurs Educ Perspect. 2005 Mar-Apr;26(2):96-103. PMID 15921126
- [Result] Hopewell S, Chan AW, Collins GS, Hrobjartsson A, Moher D, Schulz KF, Tunn R, Aggarwal R, Berkwits M, Berlin JA, Bhandari N, Butcher NJ, Campbell MK, Chidebe RCW, Elbourne D, Farmer A, Fergusson DA, Golub RM, Goodman SN, Hoffmann TC, Ioannidis JPA, Kahan BC, Knowles RL, Lamb SE, Lewis S, Loder E, Offringa M, Ravaud P, Richards DP, Rockhold FW, Schriger DL, Siegfried NL, Staniszewska S, Taylor RS, Thabane L, Torgerson D, Vohra S, White IR, Boutron I. CONSORT 2025 statement: updated guideline for reporting randomised trials. BMJ. 2025 Apr 14;389:e081123. doi: 10.1136/bmj-2024-081123. PMID 40228833
- [Result] Holland, K. (2019). An introduction to the Roper-Logan-Tierney model for nursing, based on Activities of Living. In K. Holland & J. Jenkins (Eds.), Applying the Roper-Logan-Tierney model in practice (3rd ed., pp. 17-39). China: Elsevier. https://doi.org/10.1016/B978-0-7020-4658-2.00002-8
- [Result] Hoang, C., Copnell, B., Lawrence, K., & Peddle, M. (2022). Undergraduate nursing education and end-of-life simulation: A scoping review. Clinical Simulation in Nursing, 70, 56-73. https://doi.org/10.1016/j.ecns.2022.06.009
- [Result] Esin, M. N. (2020). Data collection methods and tools & reliability and validity of data collection instruments. In S. Erdoğan, N. Nahcivan, & M. N. Esin (Eds.), Research in nursing: Process, application, and critique (pp. 193-232). Nobel Tıp Kitabevleri.
- [Result] Dickerson, K., Gantt, L. T., & Swanson, M. (2023). Unexpected death of a mannequin: a mixed methods pilot study on relationships of stress, anxiety, and resilience on learning outcomes. Clinical Simulation in Nursing, 74, 65-71.
- [Result] Cekic Y, Caliskan BB, Kucuk Ozturk G, Kaya Meral D, Bag B. "It was the first time someone had died before my eyes...": A qualitative study on the first death experiences of nursing students. Nurse Educ Today. 2024 Feb;133:106075. doi: 10.1016/j.nedt.2023.106075. Epub 2023 Dec 18. PMID 38134812
- [Result] Çakmak, B. (2022). The effect of repeated standardized patient-based education on knowledge, attitudes toward patients in the dying process, and emotional states of nursing students in end-of-life care (Doctoral dissertation, Ankara Yıldırım Beyazıt University, Institute of Health Sciences).
- [Result] Çakır, G. N. (2024). The effect of using two different simulation techniques in kangaroo care education during birth on the knowledge, skills, satisfaction, and self-confidence levels of nursing students: A randomized controlled study (Master's thesis, Yeditepe University, Institute of Health Sciences). İstanbul
- [Result] Conley CE. Student nurses' end-of-life and post mortem care self-efficacy: A descriptive study. Nurse Educ Today. 2023 Feb;121:105698. doi: 10.1016/j.nedt.2022.105698. Epub 2022 Dec 17. PMID 36549255
- [Result] Ayvaz, M. Y., Dedeoğlu Demir, B., Türen, S., & Enç, N. (2021). End-of-life care in intensive care patients. In N. Enç (Ed.), Intensive care nursing (1st ed., Chapter 19, pp. 553-573). İstanbul: Nobel Tıp Kitabevleri.

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2025-08-12): https://cdn.clinicaltrials.gov/large-docs/56/NCT07125456/Prot_SAP_ICF_000.pdf